CLINICAL TRIAL: NCT03774797
Title: Immediate Postpartum LARC Implementation: Pilot Study at Michigan Medicine
Brief Title: Feasibility of Immediate Postpartum Long-acting Reversible Contraception Implementation
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle H. Moniz, Assistant Professor, University of Michigan
Other Study IDs: HUM00126810
Record Dates: First submitted 2018-11-20; First posted 2018-12-13 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy Related
Keywords: contraception; long-acting reversible contraception; postpartum; toolkit; implementation; feasibility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-Implementation Patients: Enrolled patients will take online surveys following a prenatal or a postpartum visit.
- Post-Implementation Patients: All enrolled patients will take online surveys following a prenatal or a postpartum visit. A subset will be interviewed after the postpartum survey.
  Interventions: Other: Implementation Toolkit
- Post-Implementation Providers: All enrolled providers will take online surveys at 6-12 months after program implementation, and a subset will be interviewed.
  Interventions: Other: Implementation Toolkit

INTERVENTIONS:
Other: Implementation Toolkit — Post-implementation patients and providers will be assessed after the implementation toolkit has been used to improve service delivery at the study site.
  Groups: Post-Implementation Patients; Post-Implementation Providers

SUMMARY:
The objective of this study is to test and disseminate tools that drive successful immediate postpartum Long-Acting Reversible Contraception (LARC) implementation. The long-term goal is to reduce unintended pregnancy soon after childbirth by increasing access to immediate postpartum LARC for women who desire it.

DETAILED DESCRIPTION:
Based on previous work, the investigators have generated a toolkit to guide the integration of immediate postpartum LARC services into widespread clinical practice. In the proposed work, this toolkit will be used to initiate immediate postpartum LARC services in a single site with low baseline immediate postpartum LARC uptake (Michigan Medicine). The investigators will conduct a feasibility study using mixed methods to assess acceptability and appropriateness of toolkit items; patient experience of care; immediate postpartum LARC utilization rate; and prenatal contraceptive counseling rate.

ELIGIBILITY:
Inclusion Criteria:

* Female (patients)
* Pregnant (patients)
* Receiving obstetrical care at Michigan Medicine (patients)
* L&D provider at Michigan Medicine (providers)

Exclusion Criteria:

* non-English speaking
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes women receiving prenatal care and maternity providers working at the study site. The patient populations includes approximately 5000 women annually. The provider population includes approximately 400 maternity providers.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-08-16 (Actual)

PRIMARY OUTCOMES:
Patient experience of care | Surveys will be collected from pregnant or postpartum women, during the 6-12 months after implementation of a new protocol for peripartum contraceptive care
  Patient online surveys about their experience of care during prenatal visits, hospital stay, or postpartum office visit
Acceptability of care process - patients | Surveys will be collected from pregnant or postpartum women, during the 6-12 months after implementation of a new protocol for peripartum contraceptive care
  Online survey assessing experience of care, acceptability and appropriateness of implementation tools
Appropriateness of care process - patients | Surveys will be collected from pregnant or postpartum women, during the 6-12 months after implementation of a new protocol for peripartum contraceptive care
  Online survey assessing experience of care, acceptability and appropriateness of implementation tools
Acceptability of implementation process - study site maternity care providers | Surveys will be collected during the 6-12 months after implementation of a new protocol for peripartum contraceptive care
  Online survey assessing overall experience of care delivery, acceptability and appropriateness of implementation tools
Appropriateness of implementation process - study site maternity care providers | Surveys will be collected during the 6-12 months after implementation of a new protocol for peripartum contraceptive care
  Online survey assessing overall experience of care delivery, acceptability and appropriateness of implementation tools

SECONDARY OUTCOMES:
Acceptability of implementation toolkit items - patients | Interviews will take place after the survey is completed, during the 6-18 months after implementation of a new protocol for peripartum contraceptive care
  30-minute follow-up in-person interview of subgroup of patients who completed surveys
Appropriateness of implementation toolkit items - patients | Interviews will take place after the survey is completed, during the 6-18 months after implementation of a new protocol for peripartum contraceptive care
  30-minute follow-up in-person interview of subgroup of patients who completed surveys
Acceptability of implementation toolkit items - providers | Interviews will take place after the survey is completed, during the 6-18 months after implementation of a new protocol for peripartum contraceptive care
  30-minute follow-up in-person interview of subgroup of providers who completed survey
Appropriateness of implementation toolkit items - providers | Interviews will take place after the survey is completed, during the 6-18 months after implementation of a new protocol for peripartum contraceptive care
  30-minute follow-up in-person interview of subgroup of providers who completed survey
Perinatal contraceptive counseling rate | Measured monthly, up to 24 months after toolkit implementation
  Proportion of delivered patients with documentation of prenatal counseling about postpartum contraception
Immediate postpartum LARC provision rate | Measured monthly, up to 24 months after toolkit implementation
  Proportion of delivered patients with documentation of preference for immediate postpartum LARC who receive a LARC device

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H. Moniz, MD, MSc, Principal Investigator — University of Michigan; Vanessa K. Dalton, MD, MPH, Principal Investigator — University of Michigan; Michelle Heisler, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States